CLINICAL TRIAL: NCT03741179
Title: A Phase III, Multicentric, Randomized, Open-label, Parallel-group Clinical Trial to Detect False Positives From First-trimester Preeclampsia Screening (StopPRE) at the Second-trimester of Pregnancy
Brief Title: Detection of False Positives From First-trimester Preeclampsia Screening (StopPRE) at the Second-trimester of Pregnancy
Acronym: StopPRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOPPRE; 2018-000811-26 (EudraCT Number)
Record Dates: First submitted 2018-10-25; First posted 2018-11-14 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Pre-Eclampsia
Keywords: pre-eclampsia; pregnant; sFlt-1/PlGF ratio; ASA treatment
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: A phase III, multicentric, Randomized, open-label, parallel-group clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASA-withdrawn group (Experimental): ASA treatment will be withdrawn if patients present an sFlt/PlGF < 38 at 24+0-27+6 weeks of gestation.
  Interventions: Drug: ASA-withdrawn group
- ASA group (No Intervention): ASA treatment will continue until 36 weeks of gestation if patients present an sFlt/PlGF ratio < 38 at 24+0-27+6 weeks of gestation.

INTERVENTIONS:
Drug: ASA-withdrawn group — Patients whith sFlt/PlGF ratio < 38 at 24+0-27+6 weeks will be randomized into two arms of the trial. Patients allocated in the experimental arm will stop the ASA treatment.
  Other Names: sFlt y PlGF ratio less than 38.
  Arms: ASA-withdrawn group

SUMMARY:
Pregnant women at a higher risk for pre-eclampsia (PE) should be offered preventive daily treatment with acetylsalicylic acid (ASA) started before 16 weeks of gestation. To select patients at higher risk for PE, multiparametric assessment combining maternal history, biochemical factors and biophysical factors should be used during the first trimester of pregnancy. Multiparametric risk assessments have a detection rate for early-onset PE around 80% at a false positive rate of 10%. Owing to the low prevalence of early-onset and preterm PE, more than 90% of patients considered at high risk, at the first-trimester screening, will not eventually develop PE. Thus, ASA treatment would be innecessary and could be safely discontinued in these patients.

The sFlt-1 to PlGF ratio has a high negative predictive value for PE during the second and third trimester of pregnancy. Thus, it could be used to detect false-positive patients from the first-trimester screening.

This is a multicentric, randomized, open, parallel, controlled, phase III trial, where 1,080 patients under treatment with ASA for being at high risk for preeclampsia from the first-trimester screening, will be candidates to participate. Patients with a sFlt-1/PlGF <38, from 24 to 27+6 weeks of gestation will be randomized at a 1:1 ratio and allocated to either continue ASA until 36 weeks or to stop ASA treatment.

DETAILED DESCRIPTION:
The main objective of the study is to demonstrate that in patients considered to be at high risk for PE (from the first-trimester screening) and with sFlt-1/PlGF ratio <38, between 24+0 and 27+6 weeks, the incidence of preterm PE, after cessation of the treatment with ASA, will not be superior to that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Gestational age between 24+0 and 27+6 weeks
* Single pregnancy
* High-risk for pre-eclampsia from the first-trimester screening for pre-eclampsia
* ASA treatment started before or at 16+6 weeks of gestation
* Maternal sFlt-1/PlGF ratio at 24+0-27+6 weeks of gestation
* Signed informed consent

Exclusion Criteria:

* Multiple pregnancy
* Dead and/or fetal polymalformation, including also any fetal genetical and/or chromosomic disease.
* Von Willebrand disease.
* ASA intolerance and /or allergy
* Peptic ulcer
* ASA compliance <50% before inclusion
* Patients with misunderstanding or not able to understand the protocol, including also any condition which could compromise the compliance of the protocol, according to the investigator's opinion.
* No signature of the informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of preterm pre-eclampsia in both arms of the study (ASA vs no ASA). | From 24+0 weeks of gestation onwards
  Rate of pre-eclampsia <37 weeks in pregnant women at high-risk for early-onset PE from the first-trimester screening and ratio sFlt-1/PlGF<38 between 24-27+6 weeks of gestation in both arms of the study (ASA vs no ASA).

CONTACTS AND LOCATIONS:
Overall Officials: Manel Mendoza Cobaleda, MD, PhD, Principal Investigator — Vall d'Hebron Institut de Recerca (VHIR)
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Derived] Mendoza M, Bonacina E, Garcia-Manau P, Lopez M, Caamina S, Vives A, Lopez-Quesada E, Ricart M, Maroto A, de Mingo L, Pintado E, Ferrer-Costa R, Martin L, Rodriguez-Zurita A, Garcia E, Pallarols M, Vidal-Sagnier L, Teixidor M, Orizales-Lago C, Perez-Gomez A, Ocana V, Puerto L, Millan P, Alsius M, Diaz S, Maiz N, Carreras E, Suy A. Aspirin Discontinuation at 24 to 28 Weeks' Gestation in Pregnancies at High Risk of Preterm Preeclampsia: A Randomized Clinical Trial. JAMA. 2023 Feb 21;329(7):542-550. doi: 10.1001/jama.2023.0691. PMID 36809321